CLINICAL TRIAL: NCT04872296
Title: Early Weight Bearing for Isolated Fibular Fractures: A Prospective Randomized Study
Brief Title: Weight Bearing for Fibular Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RSHA18D.798
Record Dates: First submitted 2021-05-03; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Fibula Fracture
MeSH Terms: conditions — Fibula Fractures | interventions — Complementary Therapies; Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early weight bearing (Active Comparator): Participants treated for an ankle fracture will be allowed to weight bear early after surgery starting at 2 weeks post operatively
  Interventions: Device: Controlled Ankle Motion (CAM) boot; Procedure: Physical Therapy
- Postponed weight bearing (Active Comparator): Participants treated for an ankle fracture will be treated with standard protocol of non-weight bearing for 6 weeks post operatively.
  Interventions: Device: Controlled Ankle Motion (CAM) boot; Procedure: Physical Therapy

INTERVENTIONS:
Device: Controlled Ankle Motion (CAM) boot — A CAM boot will be worn on the affected ankle to allow weight bearing
Procedure: Physical Therapy — Standard physical therapy protocol will be started at 6 weeks after surgery

SUMMARY:
It is common practice to restrict weight bearing after ankle fracture open reduction and internal fixation (ORIF) until week 6 postoperatively. However, controversy exists surrounding the optimal postoperative protocol. At our institution, all ankle fractures are made non-weight bearing for 6 weeks across the board. Isolated lateral malleolar fractures after ORIF may benefit from earlier weight bearing in terms of patient satisfaction, short-term functionality, and return to work. The purpose of this study is to determine if early weight bearing at 2 weeks postoperatively for isolated lateral malleolar fractures leads to a higher satisfaction with surgery as compared to standard protocol for postoperative ankle fractures and better functional outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age>18) undergoing surgical treatment for isolated lateral malleolar fracture with foot and ankle surgeons at the Rothman Orthopaedic Institute

Exclusion Criteria:

* Patients requiring other fracture fixation, deltoid ligament repair, or syndesmosis fixation
* Revision ankle fracture cases
* Pre-existing impaired mobility,
* Pre-existing cognitive disability,
* Open fractures,
* BMI >40,
* Diabetes mellitus (DM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Participant Satisfaction with treatment #1 | 24 weeks
  Participant satisfaction will be measured using the Short Form-12 survey (SF-12)
Participant Satisfaction with treatment #2 | 24 weeks
  Participant satisfaction will be measured using the Foot and Ankle Ability Measure (FAAM) scores
Participant Pain after surgery | 24 weeks
  Participant Pain will be measured using the Visual Analog Scale for Pain (VAS) score

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States